CLINICAL TRIAL: NCT00044616
Title: Relapse Prevention of Bipolar Type-II Disorder
Brief Title: Relapse Prevention for Bipolar Type-II Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH060353-01 (NIH); R01MH060353-01 (NIH); DSIR 83-ATP
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2013-12

CONDITIONS: Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Fluoxetine; Lithium

INTERVENTIONS:
Drug: Fluoxetine
Drug: Lithium

SUMMARY:
This 62-week study will compare the safety and effectiveness of fluoxetine (Prozac®), lithium, the combination of these two medications, and placebo in treating and preventing recurrent depressive episodes in people with bipolar type II disorder.

DETAILED DESCRIPTION:
Bipolar II (BP II) disorder is characterized by a high recurrence of major depressive episodes (MDE), and it is associated with substantial illness and deaths. Unfortunately, relatively little attention has been given to treatment of BP II. Concern that patients may switch from depressed to manic states during treatment of MDE has impeded the development of effective treatments for BP II MDE.

BP II MDE patients are treated initially with fluoxetine for 10 weeks. Patients who recover from MDE are then randomized to receive a relapse-prevention treatment of fluoxetine, lithium, a combination of fluoxetine and lithium, or placebo for 1 year. Patients undergo clinical and laboratory evaluations, including physical examinations, bloodwork, thyroid function tests, electrocardiogram (ECG), urinalysis, and HAM-D, YMR, CGI-S, CGI-I, and adverse events scales.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00602537

ELIGIBILITY:
Inclusion Criteria:

* Bipolar II Depression

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2001-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Depression Research Unit, Univ Penn, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Amsterdam JD, Luo L, Shults J. Efficacy and mood conversion rate during long-term fluoxetine v. lithium monotherapy in rapid- and non-rapid-cycling bipolar II disorder. Br J Psychiatry. 2013 Apr;202(4):301-6. doi: 10.1192/bjp.bp.111.104711. Epub 2012 Oct 25. PMID 23099447
- [Derived] Amsterdam JD, Shults J. Efficacy and safety of long-term fluoxetine versus lithium monotherapy of bipolar II disorder: a randomized, double-blind, placebo-substitution study. Am J Psychiatry. 2010 Jul;167(7):792-800. doi: 10.1176/appi.ajp.2009.09020284. Epub 2010 Apr 1. PMID 20360317